CLINICAL TRIAL: NCT01820117
Title: Brain Integrity in Survivors of Hodgkin Lymphoma (HL) Treated With Thoracic Radiation
Brief Title: Brain Integrity in Survivors of Hodgkin Lymphoma Treated With Thoracic Radiation
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: BRIGHT; R01CA174794 (NIH)
Record Dates: First submitted 2013-03-21; First posted 2013-03-28 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Hodgkin Lymphoma
Keywords: long-term health outcomes
MeSH Terms: conditions — Hodgkin Disease | interventions — Patient Health Questionnaire; Exercise Test; Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood (5 ml) will be collected, frozen and stored for future serum biomarker assays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hodgkin lymphoma: Participants previously treated at St. Jude Children's Research Hospital with thoracic radiation therapy for Hodgkin lymphoma.
  Interventions: Neurocognitive Evaluation, Quantitative Brain Imaging, Neurologic Evaluation, Comprehensive Health Questionnaire, Vascular Testing, Cardiopulmonary Exercise Testing, Echocardiography, Pulmonary Function Testing, Serum Biomarkers, and Ophthalmology Examination.
  Interventions: Other: Neurocognitive Evaluation; Other: Quantitative Brain Imaging; Other: Neurologic Evaluation; Other: Health Questionnaire; Other: Vascular Testing; Other: Cardiopulmonary Exercise Testing; Other: Echocardiography; Other: Pulmonary Function Testing; Procedure: Serum Biomarkers; Other: Ophthalmology Examination
- Normal control: A group of healthy individuals matched for age, sex and race.
  Interventions: Neurocognitive Evaluation, Quantitative Brain Imaging, Neurologic Evaluation, Comprehensive Health Questionnaire, Vascular Testing, Cardiopulmonary Exercise Testing, Echocardiography, Pulmonary Function Testing, Serum Biomarkers, and Ophthalmology Examination.
  Interventions: Other: Neurocognitive Evaluation; Other: Quantitative Brain Imaging; Other: Neurologic Evaluation; Other: Health Questionnaire; Other: Vascular Testing; Other: Cardiopulmonary Exercise Testing; Other: Echocardiography; Other: Pulmonary Function Testing; Procedure: Serum Biomarkers; Other: Ophthalmology Examination

INTERVENTIONS:
Other: Neurocognitive Evaluation — The neurocognitive evaluation will include measures of academic achievement, intelligence, sustained attention, memory, processing speed, executive functions, functional behavior, and emotional functioning.
Other: Quantitative Brain Imaging — Imaging will include raw images to both quantify white matter hyperintensities and hemosiderin deposits, as well as cortical thickness and tissue segmentation. Brain imaging will be repeated on participants who are concurrently enrolled on BRIGHT and MIND protocols at St. Jude and who completed prior brain imaging during the BRIGHT clinic visit. The repeat MRI will be done at their 6 month MIND clinic visit.
Other: Neurologic Evaluation — Evaluation includes a complete review of neurologic symptoms, and interview and examination by the neurologist, assessment of neurologic symptoms and determination of their impact on day-to-day living, and quantified neurologic examination by the neurologist.
Other: Health Questionnaire — Participants will be asked to complete an approximately 450-item survey to assess health history and status, social and demographic factors, health behaviors, and psychosocial constructs.
Other: Vascular Testing — Digital assessment of endothelial function will be studied, and central blood and pulse pressure and carotid-femoral pulse wave velocity will be non-invasively measured.
Other: Cardiopulmonary Exercise Testing — Study participants will undergo cardiopulmonary exercise testing by treadmill. Those participants whose physical performance does not permit walking safely on the treadmill (extreme deconditioning, lower extremity paralysis, balance disorder, acute lower extremity injury) will perform cardiopulmonary exercise testing on a bicycle or upper extremity ergometer using a comparable testing protocol.
Other: Echocardiography — A complete 3D as well as 2D echocardiogram with Doppler and M-mode will be performed.
Other: Pulmonary Function Testing — Pulmonary function testing will include spirometry, lung volume measurements by body plethysmography, and single-breath carbon monoxide-diffusion capacity (DLCO).
Procedure: Serum Biomarkers — Blood for serum biomarkers associated with cardiovascular morbidity will be drawn, including high-sensitivity C-reactive protein, serum homocysteine.
Other: Ophthalmology Examination — Ophthalmology examination will include a review of symptoms, examination, and fundus imaging. The examination will consist of visual acuity testing, refraction testing, retinoscopy, ocular pressure, and examination under mydriasis. Fundus photography will be used to capture an image of the retina for examination of potential hypertensive retinopathy.

SUMMARY:
While thoracic radiation therapy (TRT) has been a primary component in successful treatment of a variety of childhood and adult cancers, the exposure to this treatment has been associated with significant cardiovascular and pulmonary morbidity in long-term survivors. Within non-cancer populations, cardiovascular and pulmonary morbidity is associated with increased risk for cerebral vascular accidents (CVAs), accelerated brain atrophy and neurocognitive impairment. Patients with chronic heart disease demonstrate problems with attention, processing speed, memory, and executive functions. Chronic pulmonary disease also increases the risk of stroke, leukoencephalopathy, and neurocognitive impairment in non-cancer populations. The investigators propose to examine indices of brain integrity, including neurocognitive performance and brain MRI/MRA, in long-term adult survivors of Hodgkin lymphoma (HL) treated with thoracic radiation and no direct central nervous system therapy.

OBJECTIVES:

1. To evaluate brain integrity in adult survivors of childhood HL treated with thoracic radiation therapy.
2. To identify therapeutic factors associated with brain integrity in adult survivors of childhood HL who are at risk for cardiac and pulmonary morbidity.
3. To examine associations between cardiac, vascular and pulmonary health and brain integrity in adult survivors of childhood HL treated with thoracic radiation.

DETAILED DESCRIPTION:
This is an observational study to collect health data from long-term survivors of Hodgkin lymphoma (HL). Data will be collected once at participant enrollment. The long-term effects of thoracic radiation therapy (TRT) given earlier as part of the treatment for HL will be examined in long-term survivors and compared to health data collected from normal volunteers.

HL survivors who were treated at St. Jude Children's Research Hospital (SJCRH) with TRT will be recruited to complete a comprehensive neurocognitive evaluation, brain MRI/MRA, a clinical neurological exam, peripheral pulse contour analysis, non-invasive central blood pressure monitoring, cardiopulmonary exercise testing, and serum biomarkers related to cardiac disease. As part of their standard St. Jude LIFE protocol evaluation, they also complete an echocardiogram, pulmonary function tests and questionnaires designed to evaluate broad health, psychological, socioeconomic and environmental factors that impact everyday life.

A comparison sample of healthy individuals, frequency-matched on age, sex and race will also be recruited. The comparison group will complete the comprehensive neurocognitive evaluation, brain MRI/MRA, clinical neurological exam, pulse contour analysis, non-invasive central blood pressure monitoring, and cardiopulmonary exercise testing. Through the St. Jude LIFE protocol, the comparison sample will also complete an echocardiogram, pulmonary function tests and questionnaires designed to evaluate broad health, psychological, socioeconomic and environmental factors that impact everyday life.

ELIGIBILITY:
Inclusion Criteria - HL participant:

* Current St. Jude LIFE protocol Participant, treated with thoracic radiation
* Currently ≥ 18 years of age
* ≥ 10 years from original diagnosis

Exclusion Criteria - HL participant:

* Has participated in the previous pilot study at St. Jude (HPP16)
* History of cranial or total-body radiation therapy
* History of intrathecal Methotrexate, high-dose Methotrexate or high-dose Cytarabine.
* History of head injury or diagnosis of a genetic disorder associated with neurocognitive impairment
* Pre-existing known neurocognitive impairment prior to diagnosis of Hodgkin lymphoma
* History of congenital heart disease reported in the literature to be associated with neurocognitive status as determined by the principal investigators
* Currently pregnant
* Secondary central nervous system neoplasm

Inclusion Criteria - Normal Control:

* Research participant is a sibling, parent, relative or friend of a current or former St. Jude patient
* Research participant must be at least 18 years of age at the time of the scheduled evaluation

Exclusion Criteria - Normal Control:

* History of cranial, total-body or thoracic radiation therapy
* History of intrathecal Methotrexate, high-dose Methotrexate, or high-dose Cytarabine.
* History of head injury or diagnosis of a genetic disorder associated with neurocognitive impairment
* Known neurocognitive impairment
* History of congenital heart disease reported in the literature to be associated with neurocognitive status as determined by the principal investigators
* Currently pregnant
* Central nervous system neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SJLIFE is an institutional initiative to establish a lifetime survivor cohort to study physical and behavioral health outcomes in adult survivors of childhood cancer. This protocol includes individuals diagnosed and treated with a malignancy during childhood at SJCRH since 1962, who are now 10 or more years from diagnosis and over 18 years of age.
  The current study will recruit participants from the SJLIFE cohort who received thoracic radiation as part of their treatment for Hodgkin lymphoma.
  Potentially eligible comparison group participants will be recruited from the relative or friend population who accompany any After Completion of Therapy (ACT) or SJLIFE patient for follow-up at SJCRH.
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2013-04-26 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Neurocognitive measures of sustained attention and memory between HL survivor group and control group. | Once, at or near enrollment
  To evaluate brain integrity in adult survivors of childhood cancer treated with thoracic radiation therapy.
  Two-sided two-sample t test will be conducted to compare the difference of neurocognitive impairment in area of sustained attention and memory in the HL survivors and matched controls.
Rate of leukoencephalopathy and hemosiderin deposits on quantitative MRI between HL survivor group and control group. | Once, at or near enrollment
  To evaluate brain integrity in adult survivors of childhood cancer treated with thoracic radiation therapy.
  Two-sided two-sample proportional test will be used to compare the rates of leukoencephalopathy and hemosiderin deposits between in the HL survivors and matched controls.
Rate of neurologic symptoms between HL survivor group and control group. | Once, at or near enrollment
  To evaluate brain integrity in adult survivors of childhood cancer treated with thoracic radiation therapy.
  Two-sided two-sample proportional test will be used to compare the rates of neurologic symptoms between the HL survivors and matched controls.

SECONDARY OUTCOMES:
Association between thoracic radiation dose and sustained attention and memory scores and rate of leukoencephalopathy and hemosiderin deposits in HL survivors. | Once, at or near enrollment
  In HL survivors only, outcome variables will be: sustained attention (continuous), memory (continuous), leukoencephalopathy (dichotomous) and hemosiderin deposits (dichotomous). Independent variables are radiation dose to cardiopulmonary structures. Covariates will include chemotherapy exposures, particularly anthracycline exposure. For each continuous response variable, linear regression model will be used to see its association with these independent variables, adjusted for race/age/sex. Other possible covariates include educational attainment, employment and occupation, current physical activity, and alcohol and tobacco. For each dichotomous response variable, logistic regression model will be used to see its association with these independent variables, adjusted for race/age/sex. AIC criteria will be used to select the final model.
Association between cardiac, vascular and pulmonary health and sustained attention and memory scores and rate of leukoencephalopathy and hemosiderin deposits. | Once, at or near enrollment
  In HL survivors only, outcome variables will be: sustained attention (continuous), memory (continuous), leukoencephalopathy (dichotomous) and hemosiderin deposits (dichotomous). Independent variables are cardiac, vascular and pulmonary health. For each continuous response variable, linear regression model will be used to see its association with these independent variables, adjusted for race/age/sex. Other possible covariates include educational attainment, employment and occupation, current physical activity, and alcohol and tobacco. For each dichotomous response variable, logistic regression model will be used to see its association with these independent variables, adjusted for race/age/sex. AIC criteria will be used to select the final model.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Krull, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols